CLINICAL TRIAL: NCT05052684
Title: The Leaflex™ Brazilian Standalone Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reprioritization of attention and resources by Sponsor
Sponsor: Pi-cardia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02-CLN-019(BR)
Record Dates: First submitted 2021-09-09; First posted 2021-09-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leaflex™ Performer (Experimental): Intervention with Leaflex™ Performer
  Interventions: Device: Leaflex™ Performer

INTERVENTIONS:
Device: Leaflex™ Performer — A transfemoral catheter designed to treat calcific aortic stenosis by scoring the calcification in the aortic valve leaflets.

SUMMARY:
A prospective, multicenter, single-arm study aimed to demonstrate safety and performance of the Leaflex™ Performer in the treatment of symptomatic severe aortic stenosis.

DETAILED DESCRIPTION:
A prospective, multicenter, single-arm study aimed to demonstrate safety and performance of the Leaflex™ Performer in the treatment of symptomatic severe aortic stenosis.

Subjects will be seen at pre- and post procedure, discharge, 30 days and at 3, 6, 9 and 12 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptomatic, severe aortic stenosis who are not recommended by the heart team for immediate treatment with surgical or transcatheter aortic valve replacement.
* Patient is willing to comply with scheduled visits and tests and is able and willing to provide informed consent.

Exclusion Criteria:

* Severe aortic regurgitation.
* Anatomic contraindications.
* Coronary, carotid, or vertebral artery disease that, in the opinion of the heart team, should be treated; or treatment of coronary artery disease ≤ 1 month prior to index procedure.
* Aortic balloon valvuloplasty ≤ 3 months prior to index procedure.
* Stroke ≤ 12 months prior to index procedure.
* History of a myocardial infarction ≤ 6 weeks prior to index procedure.
* Patients with clinically significant abnormality in cell blood count, history of bleeding diathesis or coagulopathy.
* Hemodynamic instability.
* Hypertrophic cardiomyopathy with obstruction.
* Left ventricle ejection fraction <30%.
* Ongoing severe infection, including endocarditis, or sepsis.
* Life expectancy ≤ 12 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Change in aortic valve area | Baseline and up to 3 days post procedure
  Assessed by echo Assessed by echo

SECONDARY OUTCOMES:
Rate of all-cause mortality and all-cause stroke (VARC 2) | 30 days post procedure
  Composite
Rate of worsening of aortic regurgitation | Baseline and 30 days post procedure
  By more than 1 grade
Rate of device related adverse events | Up to 12 months post procedure
  Percent of patients with device related adverse events
Change in 6 minute walk test | Baseline, 1, 6 and 12 months post procedure
  Distance (meters)
Change in Quality of Life - KCCQ | Baseline, 1, 6 and 12 months post procedure
  Kansas City Cardiomyopathy Questionnaire (KCCQ)
Change in Quality of Life - EQ5D | Baseline, 1, 6 and 12 months post procedure
  EuroQol- 5 Dimension (EQ5D)
Change in aortic valve area | Baseline, up to 3 days, 30 days, 3, 6, 9 and 12 months post procedure
  Assessed by echo
Change in pressure gradients | Baseline, up to 3 days, 30 days, 3, 6, 9 and 12 months post procedure
  Assessed by echo
Change in pressure gradients | Pre-treatment, immediately post treatment (during procedure)
  Measured invasively

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Givon, Study Director — Pi-cardia
Locations (1):
- Instituto do Coração FMUSP Centro de Pesquisa, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No